CLINICAL TRIAL: NCT03310788
Title: Monitoring of the Intraocular Pressure After Selective Laser Trabeculoplasty Using iCare Home
Brief Title: Monitoring of the IOP After SLT Using iCare Home
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Erik Eye Hospital (Other)
Responsible Party: Principal Investigator, Enping Chen, MD Ph D, St. Erik Eye Hospital
Other Study IDs: HOME SLT
Record Dates: First submitted 2017-10-02; First posted 2017-10-16 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Glaucoma Open-Angle Primary; Pseudo Exfoliation Syndrome
Keywords: IOP fluctuations; iCare Home; SLT; self-tonometry
MeSH Terms: conditions — Glaucoma, Open-Angle; Exfoliation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate how much selective trabeculoplasty (SLT) influences intraocular pressure (IOP) fluctuations measured with iCare Home rebound tonometry (RTHome) in patients with primary open-angle glaucoma (POAG) or pseudo-exfoliation glaucoma (PEX).

DETAILED DESCRIPTION:
Sixty glaucoma patients (POAG and PEX) planned for SLT will be recruited.

At baseline, patients will be trained to use the iCare Home tonometer, a handheld device based on rebound tonometry and designed for patients to use at home. After the training session and when patients feel confident, a measurement will be recorded. Thereafter, a new measurement will be obtained by the study staff (an optometrist or a nurse) using the same device. No IOP values will be visible for the examiner at that point. Thereafter, a single IOP measurement will be obtained by the same study staff using Goldmann applanation tonometry (GAT). Patients will then borrow the iCare Home tonometer to meaure their IOP at 06 and 10 am, and at 2, 6 and 10 pm during three consecutive days to obtain an IOP curve. Patients will come for a second visit where new measurements will be made in the same way as at baseline.

Two months after SLT, a new IOP curve will be obtained following the same procedure as pre-operatively. Patients' daily activities (diet, motion or sleeping habits) will not be controlled.

ELIGIBILITY:
Inclusion Criteria:

* POAG
* PXG

Exclusion Criteria:

* previous SLT
* reduced hand and arm mobility (e.g. due to rheumatism)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive male and female patients, older than 18 y.o., at St Erik's Eye Hospital in Stockholm, Sweden, diagnosed with POAG or PXG and listed for a SLT.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-10-03 (Actual); Primary Completion 2022-03-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Lowering of IOP fluctuations after SLT | 2 months
  The amplitude of the IOP fluctuations pre- and post SLT will be compared

SECONDARY OUTCOMES:
Lowering of IOP level after SLT | 2 months
  Mean IOP pre- and post SLT

CONTACTS AND LOCATIONS:
Overall Officials: Enping Chen, MD Ph D, Principal Investigator — St. Erik Eye Hospital
Locations (1):
- St Erik Eye Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No